CLINICAL TRIAL: NCT04256837
Title: Effect of Transcutaneous Electrical Auricular Stimulation of the Vagus Nerve in Kidney Transplant Recipients
Acronym: VNS-KTx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study expired and was not renewed with the IRB
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-0705
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Vagus Nerve Stimulation
Keywords: Vagus Nerve; Stimulation; Immune System

STUDY DESIGN:
Intervention Model Description: The objective of this pilot, feasibility study is to examine the effects of transcutaneous electrical auricular vagus nerve stimulation (VNS) in adult patients undergoing a single kidney transplant using donors who are either living or deceased.
  Kidney transplantation patients will be stratified into two groups, namely, those receiving their kidney from a living donor and those receiving their kidney from a deceased donor. Within each strata, patients will be randomized to receive either active VNS or sham VNS. VNS will be applied for 5 minutes prior to start of surgery. The device to be used for VNS will include a handheld electrical pulse generator and a pair of electrodes to be placed at the left ear for stimulation, targeting the auricular branch of the vagus nerve which innervates the skin overlying the cymba conchae of the ear canal.
Who Masked: Participant
Masking Description: A randomization schema will be generated by the BU-FIMR by study strata (recipients of a kidney from a living donor and recipients of a kidney from a deceased donor) using the method of permuted blocks. For those receiving their kidneys from living donors, subjects will be randomly assigned in a 1:1 ratio to either 'aVNS' or 'sVNS. For those receiving their kidneys from deceased donors, subjects will also be randomly assigned in a 1:1 ratio to either 'aVNS' or 'sVNS'. Details of the randomization procedure, including required record keeping will be further developed upon approval of the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VNS - Live donor kidney recipients. (Experimental): Live donor kidney recipients. VNS will be applied for 5 minutes prior to start of surgery. The device to be used for VNS will include a handheld electrical pulse generator and a pair of electrodes to be placed at the left ear for stimulation, targeting the auricular branch of the vagus nerve which innervates the skin overlying the cymba conchae of the ear canal.
  Interventions: Device: Transcutaneous electrical auricular vagus nerve stimulation (VNS)
- sham VNS - Live donor kidney recipients. (Sham Comparator): Live donor kidney recipients. As above, but without applying any VNS
  Interventions: Device: Transcutaneous electrical auricular vagus nerve stimulation (VNS)
- VNS - Deceased donor kidney recipients. (Experimental): Deceased donor kidney recipients. VNS will be applied for 5 minutes prior to start of surgery. The device to be used for VNS will include a handheld electrical pulse generator and a pair of electrodes to be placed at the left ear for stimulation, targeting the auricular branch of the vagus nerve which innervates the skin overlying the cymba conchae of the ear canal.
  Interventions: Device: Transcutaneous electrical auricular vagus nerve stimulation (VNS)
- sham VNS - Deceased donor kidney recipients. (Sham Comparator): Deceased donor kidney recipients. As above, but without applying any VNS
  Interventions: Device: Transcutaneous electrical auricular vagus nerve stimulation (VNS)

INTERVENTIONS:
Device: Transcutaneous electrical auricular vagus nerve stimulation (VNS) — Electrical auricular stimulation is accomplished using a Roscoe Medical TENS 7000 that delivers a programmable electrical current density, frequency, and pulse width. The TENS 7000 will be connected to ear clip (or hand held) electrodes to transcutaneously stimulate the cymba conchae of the ear to activate the auricular branch of the vagus nerve (diagram above), also known as Arnold's nerve, which provides sensory innervation to the skin surrounding the ear canal. Through a neural reflex arc, activation of this sensory nerve sends a neural signal to the brainstem that then activates the efferent vagus nerve through the nucleus of the solitary tract (NTS). This is a well-described and clinically accepted neuromodulatory pathway, as transcutaneous electrical auricular stimulation has been studied to treat seizures, similarly to how invasive electrical vagus nerve stimulation has been approved by the FDA for the past two decades for the same indication.

SUMMARY:
Kidney transplantation entails the implantation of a live or deceased organ into a recipient. As a result of this event, there is an inflammatory response in the recipient elicited by the transplanted organ.

At the present time, immunosuppressive treatments are routinely used to avoid rejection of the transplanted organ. Although effective in this goal, there is currently an unmet need to develop new strategies to control the innate inflammatory responses and to reduce the injury caused to the organs being transplanted.

The investigators propose a novel approach to the management of this inflammatory response. The investigators will explore the "cholinergic anti-inflammatory pathway" as a potential target, a pathway first characterized in the basic science laboratories of the Feinstein Institute for Medical Research. In short, the vagus nerve activates the splenic nerve which activates choline acetyltransferase expressing T cells in the spleen. Stimulation of the alpha7 nicotinic acetylcholine receptor (alpha7nAChR) on macrophages by acetylcholine reduces production of multiple pro-inflammatory cytokines.

Currently, vagus nerve stimulation is used to treat a number of human diseases, including epilepsy, depression and migraine headaches. Many of these treatments activate the vagus nerve non-invasively by stimulating a branch of the vagus that innervates the ear. In this study, the investigators will stimulate this branch of the vagus nerve, and look for changes in inflammatory markers in the blood of kidney transplant recipients of both live and deceased donors.

Successful completion of this study will allow for future studies in organ transplant recipients.

DETAILED DESCRIPTION:
Intervention and comparators:

Patients will receive transcutaneous stimulation of the auricular branch of the left vagus nerve for 5 minutes in the OR already under anesthesia. Subjects will be blinded to their treatment arm.

The device to be used will include a handheld electrical pulse generator and a pair of electrodes to be placed at the ear for stimulation. The specific target at the ear will be the auricular branch of the vagus nerve which innervates the skin overlying the cymba conchae of the ear canal.

Anatomical landmarks and cutaneous innervation of the external ear. Three nerves contribute to the cutaneous innervation of the lateral aspect of the ear: the auricular branch of the vagus nerve (ABVN), the auriculotemporal nerve (ATN) and the great auricular nerve (GAN). There is a variable degree of overlap in the distribution of these cutaneous nerves.

Electrodes will be placed near/at the entrance to the canal of the ear to provide stimulation to the auricular branch. The handheld electrical pulse generator (e.g. Roscoe Medical, TENS 7000) will be programmed to deliver stimulation pulses to the electrodes. The electrodes will be made of conductive material facilitating trans-cutaneous electrical stimulation. All subjects will be told that they may or may not sense the stimulation.

Attempts to diminish pain associated with blood drawing will be made by performing whenever possible the phlebotomy coincident with other blood drawing requirements or while the patient is under anesthesia.

The investigators will administer transcutaneous electrical stimulation to the left ears for 5 minutes. Subjects receiving auricular stimulation will receive stimulation using the following parameters: 0.300 milliseconds (msec) stimulus peaks at a frequency of 30 Hz for five (5) minutes, with peak current pulse amplitude set to 1.5 milliamps (mA). Research subjects will receive hemodynamic monitoring and heart rate variability monitoring while undergoing vagal stimulation as a routine part of the underlying care for organ procurement or anesthesia management.

Transcutaneous electrical stimulation Electrical auricular stimulation is accomplished using a Roscoe Medical TENS 7000 that delivers a programmable electrical current density, frequency, and pulse width. The TENS 7000 will be connected to ear clip (or hand held) electrodes to transcutaneously stimulate the cymba conchae of the ear to activate the auricular branch of the vagus nerve (diagram above), also known as Arnold's nerve, which provides sensory innervation to the skin surrounding the ear canal. Through a neural reflex arc, activation of this sensory nerve sends a neural signal to the brainstem that then activates the efferent vagus nerve through the nucleus of the solitary tract (NTS). This is a well-described and clinically accepted neuromodulatory pathway, as transcutaneous electrical auricular stimulation has been studied to treat seizures, similarly to how invasive electrical vagus nerve stimulation has been approved by the FDA for the past two decades for the same indication. Currently, transcutaneous electrical auricular stimulation is approved in Europe for the treatment of seizures.

The scientific basis for these specific choices comes from more than 10 years of experience performing experimental vagus nerve stimulation in animals to control bleeding at The Feinstein Institute for Medical Research. The frequency of stimulus peaks will be 30 Hz. The pulse width of the individual stimulus peaks will be 0.300 milliseconds (msec). The total duration of stimulation will be five (5) minutes. For the remaining stimulation parameter, which is the peak current pulse amplitude, the investigators will use 1.5 milliamps (mA). These stimulation parameters are very similar to parameters previously demonstrated to be safe in two separate tinnitus studies (6, 7). A portable, battery-powered oscilloscope will be used to confirm peak current.

Safety procedures Recent assessments of cardiac safety following transcutaneous electrical stimulation of the auricular branch of the vagus nerve have revealed no indication of arrhythmic effects of tVNS (6, 7).

In the exceedingly rare instance that a research subject develops a symptomatic bradyarrhythmia, qualified personnel anesthesiologists/surgeons/residents/CRNA) will be immediately available to administer any therapies (intravenous fluid, anti-arrhythmic medications, cardioversion) to treat the bradyarrhythmia and its associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients of both live and deceased donors

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Levels of blood inflammatory cytokines in kidney transplant recipients after transcutaneous auricular electrical vagus nerve stimulation. | 24 months
  The present study will measure systemic cytokines IL-1, IL-2, IL-4, IL-5, IL-6, IL-10, IL-12, IL-17, IL-22, IL-23, TNF, IFN-gamma, HMGB1, TGF-beta, GM-CSF, CXCL8, G-CSFas well as complement 1-9 in the blood of kidney transplant recipients who have undergone transcutaneous auricular electrical vagus nerve stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto P Molmenti, MD PhD MBA, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
Information on live and deceased donors will be limited to that provided by the UNOS ID that does not contain any PHI.

REFERENCES:
- [Background] Panebianco M, Rigby A, Weston J, Marson AG. Vagus nerve stimulation for partial seizures. Cochrane Database Syst Rev. 2015 Apr 3;2015(4):CD002896. doi: 10.1002/14651858.CD002896.pub2. PMID 25835947
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part II. Headache. 2016 Feb;56(2):259-66. doi: 10.1111/head.12650. Epub 2015 Sep 18. PMID 26381725
- [Background] Ben-Menachem E. Vagus nerve stimulation, side effects, and long-term safety. J Clin Neurophysiol. 2001 Sep;18(5):415-8. doi: 10.1097/00004691-200109000-00005. PMID 11709646
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part III. Headache. 2016 Mar;56(3):479-90. doi: 10.1111/head.12649. Epub 2015 Sep 14. PMID 26364805
- [Background] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Background] Kreuzer PM, Landgrebe M, Husser O, Resch M, Schecklmann M, Geisreiter F, Poeppl TB, Prasser SJ, Hajak G, Langguth B. Transcutaneous vagus nerve stimulation: retrospective assessment of cardiac safety in a pilot study. Front Psychiatry. 2012 Aug 7;3:70. doi: 10.3389/fpsyt.2012.00070. eCollection 2012. PMID 22891061
- [Background] Shim HJ, Kwak MY, An YH, Kim DH, Kim YJ, Kim HJ. Feasibility and Safety of Transcutaneous Vagus Nerve Stimulation Paired with Notched Music Therapy for the Treatment of Chronic Tinnitus. J Audiol Otol. 2015 Dec;19(3):159-67. doi: 10.7874/jao.2015.19.3.159. Epub 2015 Dec 18. PMID 26771015
- [Background] Huston JM, Tracey KJ. The pulse of inflammation: heart rate variability, the cholinergic anti-inflammatory pathway and implications for therapy. J Intern Med. 2011 Jan;269(1):45-53. doi: 10.1111/j.1365-2796.2010.02321.x. PMID 21158977
- [Background] Huston JM, Rosas-Ballina M, Xue X, Dowling O, Ochani K, Ochani M, Yeboah MM, Chatterjee PK, Tracey KJ, Metz CN. Cholinergic neural signals to the spleen down-regulate leukocyte trafficking via CD11b. J Immunol. 2009 Jul 1;183(1):552-9. doi: 10.4049/jimmunol.0802684. PMID 19542466
- [Background] Huston JM, Wang H, Ochani M, Ochani K, Rosas-Ballina M, Gallowitsch-Puerta M, Ashok M, Yang L, Tracey KJ, Yang H. Splenectomy protects against sepsis lethality and reduces serum HMGB1 levels. J Immunol. 2008 Sep 1;181(5):3535-9. doi: 10.4049/jimmunol.181.5.3535. PMID 18714026
- [Background] Rosas-Ballina M, Ochani M, Parrish WR, Ochani K, Harris YT, Huston JM, Chavan S, Tracey KJ. Splenic nerve is required for cholinergic antiinflammatory pathway control of TNF in endotoxemia. Proc Natl Acad Sci U S A. 2008 Aug 5;105(31):11008-13. doi: 10.1073/pnas.0803237105. Epub 2008 Jul 31. PMID 18669662
- [Background] Huston JM, Gallowitsch-Puerta M, Ochani M, Ochani K, Yuan R, Rosas-Ballina M, Ashok M, Goldstein RS, Chavan S, Pavlov VA, Metz CN, Yang H, Czura CJ, Wang H, Tracey KJ. Transcutaneous vagus nerve stimulation reduces serum high mobility group box 1 levels and improves survival in murine sepsis. Crit Care Med. 2007 Dec;35(12):2762-8. doi: 10.1097/01.CCM.0000288102.15975.BA. PMID 17901837
- [Background] Huston JM, Ochani M, Rosas-Ballina M, Liao H, Ochani K, Pavlov VA, Gallowitsch-Puerta M, Ashok M, Czura CJ, Foxwell B, Tracey KJ, Ulloa L. Splenectomy inactivates the cholinergic antiinflammatory pathway during lethal endotoxemia and polymicrobial sepsis. J Exp Med. 2006 Jul 10;203(7):1623-8. doi: 10.1084/jem.20052362. Epub 2006 Jun 19. PMID 16785311
- [Background] Rosas-Ballina M, Olofsson PS, Ochani M, Valdes-Ferrer SI, Levine YA, Reardon C, Tusche MW, Pavlov VA, Andersson U, Chavan S, Mak TW, Tracey KJ. Acetylcholine-synthesizing T cells relay neural signals in a vagus nerve circuit. Science. 2011 Oct 7;334(6052):98-101. doi: 10.1126/science.1209985. Epub 2011 Sep 15. PMID 21921156
- [Background] Wang H, Liao H, Ochani M, Justiniani M, Lin X, Yang L, Al-Abed Y, Wang H, Metz C, Miller EJ, Tracey KJ, Ulloa L. Cholinergic agonists inhibit HMGB1 release and improve survival in experimental sepsis. Nat Med. 2004 Nov;10(11):1216-21. doi: 10.1038/nm1124. Epub 2004 Oct 24. PMID 15502843
- [Background] Wang H, Yu M, Ochani M, Amella CA, Tanovic M, Susarla S, Li JH, Wang H, Yang H, Ulloa L, Al-Abed Y, Czura CJ, Tracey KJ. Nicotinic acetylcholine receptor alpha7 subunit is an essential regulator of inflammation. Nature. 2003 Jan 23;421(6921):384-8. doi: 10.1038/nature01339. Epub 2002 Dec 22. PMID 12508119
- [Background] Tracey KJ. The inflammatory reflex. Nature. 2002 Dec 19-26;420(6917):853-9. doi: 10.1038/nature01321. PMID 12490958
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541